CLINICAL TRIAL: NCT01513941
Title: Open-Label, Phase 3b Study to Determine Efficacy and Safety of Telaprevir, Pegylated-Interferon-alfa-2a and Ribavirin in Hepatitis C Virus Treatment-Naïve and Treatment-Experienced Subjects With Genotype 1 Chronic Hepatitis C and Human Immunodeficiency Virus Type 1 (HCV-1/HIV-1) Coinfection
Brief Title: An Efficacy and Safety Study of Telaprevir in Patients Infected With Both Chronic Hepatitis C Virus (HCV-1) and Human Immunodeficiency Virus (HIV-1)
Acronym: INSIGHT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR100778; VX-950HPC3008 (Other: Janssen-Cilag International NV, Belgium); 2011-004928-35 (EudraCT Number)
Record Dates: First submitted 2012-01-16; First posted 2012-01-20 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-05

CONDITIONS: Chronic Hepatitis C
Keywords: Chronic hepatitis C; Genotype 1 chronic hepatitis C; Treatment experienced with HCV-1/HIV-1 coinfection; Telaprevir; Pegylated-Interferon-alfa-2a; Ribavirin; HCV-1/HIV-1 coinfection; Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — telaprevir; Ribavirin; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Telaprevir plus Pegylated-Interferon-alfa-2a /ribavirin (RBV) (Experimental): All patients who will receive 12 weeks of treatment with telaprevir 750 mg q8h except for patients on efavirenz will receive 1125 mg every 8 hours (q8h) in combination with Pegylated-Interferon-alfa-2a (Peg-IFN-alfa-2a) 180 μg/week and RBV 800 mg/day. At Week 12, telaprevir dosing will end and the patients will continue on Peg-IFN-alfa-2a and RBV.
  Interventions: Drug: Telaprevir; Drug: Ribavirin; Drug: Pegylated-Interferon-alfa-2a

INTERVENTIONS:
Drug: Telaprevir — Type=exact number, unit=mg, number=750 or 1125, form=tablet, route=oral. the patients will receive 2 oral tablets every 8 hours for 12 weeks except for patients on efavirenz who will receive 1125mg (3 oral tablets) every 8 hours for 12 weeks.
Drug: Ribavirin — Type=exact number, unit=mg, number=400, form=tablet, route=oral. The patients will receive 2 oral ribavirin tablets twice daily for 24 or 48 weeks, based on the response guided therapy.
Drug: Pegylated-Interferon-alfa-2a — Type=exact number, unit=microgram, number=180, form=injection, route=subcutaneous The patients will receive Peg-IFN-alfa-2a 180 microgram once a week for 24 or 48 weeks; based on the response guided therapy.

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of telaprevir, given with pegylated-interferon-alfa-2a (Peg-IFN-alfa-2a) and ribavirin (RBV) in the treatment of hepatitis C in patients infected with both chronic hepatitis C virus (HCV-1) and human immunodeficiency virus (HIV-1).

DETAILED DESCRIPTION:
This is an open-label (both participant and investigator know the name of the medication given at a certain moment), single-arm, multicenter study in HCV treatment-naive and treatment-experienced patients infected with both chronic HCV-1 and HIV-1 to determine the efficacy and safety of telaprevir given with Peg-IFN-alfa-2a and RBV. The study will consist of 3 phases: a screening phase, an open-label treatment phase up to 48 weeks, and a follow-up period of 24 weeks. All patients will receive 12 weeks of treatment with telaprevir given with Peg-IFN-alfa-2a and RBV. At week 12 telaprevir dosing will end and patients will continue on Peg-IFN-alfa-2a and RBV. The total treatment duration in this study will be 24 or 48 weeks depending on the patient's prior HCV treatment status, liver disease status, and individual on-treatment virologic response in this study (equal response guided therapy). The maximum total duration of participation in the study for an individual participant will be approximately 76 weeks (screening included). Approximately 150 patients infected with both chronic HCV-1 and HIV-1 are planned to be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Chronic (detectable HCV Ribonucleic acid (RNA) more than 6 months prior screening or histological diagnosis based on liver biopsy or fibroscan) HCV infection genotype 1 with HCV RNA level greater than 1,000 IU/mL
* Confirmed diagnosis of HIV-1 infection greater than 6 months before the screening visit
* CD4 count greater than 300 cells/mm3 at screening and no value less than 200 cells/mm3 within 6 months of screening visit
* HIV-1 RNA undetectable by an ultrasensitive assay at least once within 90 days of the screening visit
* No HIV RNA values greater than 200 copies/mL within 6 months of the screening visit
* Currently taking one of the permitted anti-HIV regimens for greater than or equal to12 weeks

Exclusion Criteria:

* Anticipated need to switch anti-HIV regimen from screening through the Telaprevir treatment period
* Infection or co-infection with HCV other than genotype 1
* Contraindication to the administration of Peg-IFN-alfa or RBV
* Hepatitis B virus (HBV) co-infection
* Acute or active condition of HIV-associated opportunistic infection within 6 months of screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2012-04; Primary Completion 2014-03 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Proportion of patients achieving undetectable plasma hepatitis C virus (HCV) ribonucleic acid (RNA) levels | Up to 48 weeks
  Proportion of patients achieving sustained virologic response (SVR) undetectable plasma HCV RNA levels 12 weeks after the last planned dose of study medication.

SECONDARY OUTCOMES:
Change from baseline in log HCV RNA values | Baseline and week 48
  Change from baseline in log HCV RNA values at each time point during treatment.
Proportiond of patients achieving undetectable HCV RNA levels | Up to 48 weeks
  Proportion of patients achieving SVR24 planned, defined as having undetectable plasma HCV RNA levels 24 weeks after the last planned dose of study medication.
Proportion of patients achieving undetectable HCV RNA levels at Week 4 | Up to 48 weeks
  The proportion of patients who achieve rapid virologic response (RVR) and undetectable HCV RNA levels at Week 4 of treatment.
Proportion of patients achieving undetectable HCV RNA levels at Week 12 | Up to 48 weeks
  Proportion of patients achieving undetectable HCV RNA levels at Week 12 of treatment.
Proportion of patients achieving undetectable HCV RNA levels at Week 4 and Week 12 (eRVR) | Up to 48 weeks
  Proportion of patients achieving undetectable HCV RNA levels at Week 4 and Week 12 of treatment (eRVR).
Proportion of patients achieving undetectable HCV RNA at the actual end of treatment | Up to 48 weeks
  Proportion of patients having undetectable HCV RNA levels at the actual end of treatment (ie, Week 24, Week 48, or early discontinuation).
Proportion of patients achieving less than 25 IU/mL | Up to 48 weeks
  Proportion of patients having less than 25 IU/mL at the planned end of treatment (ie, Week 24 or Week 48).
Proportion of patients with on-treatment virologic failure | Up to 48 weeks
  Proportion of patients with on-treatment virologic failure (an increase greater than 1 log in HCV RNA level from the lowest level reached, or a value of HCV RNA greater than 100 IU/mL in patients whose HCV RNA has previously become less than 25 IU/mL during treatment).
Proportion of patients with relapse achieving detectable HCV RNA levels after previously undetectable HCV RNA levels | Up to 48 weeks
  Proportion of patients who relapse (having confirmed detectable HCV RNA during the follow-up period after previous undetectable HCV RNA levels (less than 25 IU/mL, undetectable) at planned end of treatment.
Proportion of patients with relapse achieving detectable HCV RNA levels after previous HCV RNA levels | Up to 48 weeks
  Proportion of patients who relapse, defined as having confirmed detectable HCV RNA during the follow-up period after previous HCV RNA less than 25 IU/mL at planned end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV, Belgium Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (31):
- Australia (3):
  - Cairns
  - Darlinghurst
  - Melbourne
- Brazil (4):
  - Campinas
  - Rio de Janeiro
  - Santo André
  - São Paulo
- France (4):
  - Le Kremlin-Bicêtre
  - Marseille
  - Nice
  - Paris
- Poland (3):
  - Bydgoszcz
  - Mysłowice
  - Warsaw
- Russia (5):
  - Krasnodar
  - Perm
  - Saint Petersburg
  - Smolensk
  - Voronezh
- Spain (8):
  - Alicante
  - Badalona
  - Córdoba
  - Donostia / San Sebastian
  - Elche
  - Madrid
  - Seville
  - Valencia
- Stockholm, Sweden
- United Kingdom (3):
  - Birmingham
  - Glasgow
  - London

REFERENCES:
- [Derived] Montes ML, Nelson M, Girard PM, Sasadeusz J, Horban A, Grinsztejn B, Zakharova N, Rivero A, Durant J, Ortega-Gonzalez E, Lathouwers E, Janssen K, Ouwerkerk-Mahadevan S, Witek J, Gonzalez-Garcia J. Telaprevir-based therapy in patients coinfected with chronic hepatitis C virus infection and HIV: INSIGHT study. J Antimicrob Chemother. 2016 Jan;71(1):244-50. doi: 10.1093/jac/dkv323. Epub 2015 Oct 19. PMID 26483516
- See also: Open-Label, Phase 3b Study to Determine Efficacy and Safety of Telaprevir, Pegylated- Interferon-alfa-2a and Ribavirin in Hepatitis C Virus Treatment-Naïve and Treatment-Experienced Subjects with Genotype 1 Chronic Hepatitis C and Human Immu(18137) — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=3446&filename=CR100778_CSR.pdf